CLINICAL TRIAL: NCT00451516
Title: St. John's Wort And Kava In The Treatment Of Major Depressive Disorder With Comorbid Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2006000925
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Depressive Disorder, Major; Anxiety Disorders
Keywords: Plant, medicine; Psychiatry; Major depressive disorder; Anxiety; Major Depressive Disorder with comorbid anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders | interventions — Phytotherapy; Hypericum extract LI 160

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Herbal medicine (St. John's wort and Kava)

SUMMARY:
SJW has the greatest evidence of herbal medicine efficacy in treating MDD. In treating anxiety, kava has the greatest evidence of efficacy. As comorbidity of MDD and anxiety commonly occurs, it is conceivable that a combination of an established antidepressant agent such as SJW and an established anxiolytic agent such as kava may effectively treat MDD presenting with comorbid anxiety. It is possible that a beneficial synergistic effect may also occur between SJW and kava, improving the treatment outcomes in MDD with comorbid anxiety, than by the individual substances alone. Determination of this is not addressed in this study due to limitations of time and resources. The determination of the strength of the SJW-kava combination will be ascertained by comparing similar trials using SJW and kava mono-therapy in addressing MDD and GAD.

The hypothesis is that a combination of SJW and kava will reduce MDD occurring with comorbid anxiety more than placebo.

ELIGIBILITY:
Inclusion criteria:

* Any person male or female aged 18-65 presenting with a diagnosis of unipolar depression confirmed by CIDI auto (quantified by BDI) and an anxiety score on the DASS of 8 or above i.e. the mean (quantified also by BAI)

Exclusion criteria:

* Psychotic/ Bipolar illness
* Current or < 6 month significant suicidal ideation
* Diagnosed hepato-biliary disease/inflammation
* Current or < 6 month substance abuse disorder including alcohol
* Current or < 12 month use of kava, St. John's wort,
* Current or < 1 month of synthetic antidepressants or benzodiazepines
* Previous reaction to kava or St. John's wort
* Medications that maybe pharmacokinetically altered via St. John's wort including:

  * Amitriptyline anti-coagulants e.g. phenprocoumon, warfarin,
  * Anti-fugals e.g. voriconazole,
  * Anti-histamines e.g. fexofenadine,
  * Benzodiazepines e.g. alprazolam,
  * Chemotherapeutics e.g. irinotecan, digoxin, HIV medication (anti-retrovirals), * Immunosuppressants e.g. cyclosporine, methadone, OCP,
  * Statins e.g. simvastatin, warfarin (Henderson 2002; Izzo 2004).
  * However this interactions are based on case studies and theoretical interactions and are regarded to be induced by hyperforin (a constituent of St. John's wort); low or non-standardised hyperforin preparations are regarded to not induce drug interactions as little induction of P-glycoprotein and CYP P450 enzymes occurs (Madabushi et al. 2006). Although in vitro studies have confirmed that kava and the isolated kavalactones modulate certain CYP 450 enzymes, no documented evidence of human kava-drug pharmacokinetic interactions exists (Mathews, Etheridge & Black 2002; Singh 2005)
* Seeing a psychologist or counsellor currently or in the previous month.
* Non-English speakers.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
BDI II
BAI
DASS

SECONDARY OUTCOMES:
WHOQOL
Daily Mood Monitoring Form

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Sarris, BHSc, Principal Investigator — The University of Queensland
Locations (1):
- RBWH, Brisbane, Queensland, Australia